CLINICAL TRIAL: NCT00856817
Title: Heme Oxygenase (HO) Activity and Adenosine Induced Vasodilation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment faillure. Similar study published by others. Not yet entered treatment phase.
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: P. Smits, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HOADO
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2010-01

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — Arginine; heme arginate

ARMS (2):
- 1 (Experimental): L-arginine treatment first, heme arginate treatment second
  Interventions: Drug: L-arginine + heme arginate
- 2 (Experimental): Heme arginate treatment first, L-arginine treatment second
  Interventions: Drug: Heme arginate + L-arginine

INTERVENTIONS:
Drug: L-arginine + heme arginate — L-arginine first, heme arginate second three day treatment
  Arms: 1
Drug: Heme arginate + L-arginine — Heme arginate first, L-arginine second three day treatment
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether heme oxygenase 1 induction by heme arginate treatment is of influence on adenosine induced vasodilation in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 and no older than 65 on the day of first dosing
* healthy
* Quetelet Index (Body Mass Index) of 18 to 30 kg/m2
* In general, results of haematology and chemistry should be within the laboratory's reference ranges. Determinants of renal and hepatic function should be within twice the upper limit of normal range.

Exclusion Criteria:

* Documented history of sensitivity / idiosyncrasy to medicinal products or excipients
* history of smoking within the past year
* history of or current abuse of drugs, alcohol and/or solvents
* Current use of any (over the counter) medication potentially influencing heme oxygenase or the cardiovascular system
* Inability to understand the nature and extent of the trial and the procedures required
* Participation to a drug trial within 60 days prior to the first dose
* Febrile illness within 3 days before the first dose
* Heterozygosity (LS) or homozygosity (LL) with regard to the number of GT repeats in the HO-1 promoter region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2009-03

PRIMARY OUTCOMES:
Adenosine induced vasodilation | following a three day treatment with either heme arginate or L arginine

SECONDARY OUTCOMES:
heme oxygenase expression and activity | assessed during and following a three day treatment with either heme arginate or L-arginine

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands